CLINICAL TRIAL: NCT00465010
Title: Talking Parents, Healthy Teens: A Worksite-Based Parenting Program for Parents of Adolescents
Brief Title: Effects of a Worksite Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01MH061202 (NIH)
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Adolescent Sexual Risk Behaviors
Keywords: Adolescence; Sexual health; Communication; Parenting
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Talking Parents, Healthy Teens — Talking Parents, Healthy Teens is a worksite-based parenting program to help parents of 6th-10th graders learn to promote their adolescents' healthy sexual development. The program is administered in 8 weekly one-hour sessions during the lunch hour to groups of about 15 parents and focuses on parent-adolescent relationships and communication, with an emphasis on promoting sexual health and reducing sexual risk. It is led by a trained facilitator and assistant facilitator.

SUMMARY:
Many adolescents in the U.S., even very young adolescents, are engaging in sexual risk behaviors that put them at risk for sexually transmitted diseases (STDs) and unintended pregnancy. Studies show that parents can play a significant role in promoting healthy sexual development and risk reduction among adolescents. The UCLA/RAND Center for Adolescent Health Promotion has developed Talking Parents, Healthy Teens, a worksite-based parenting program for parents of adolescents (grades 6-10) to improve parent-adolescent communication and reduce adolescent sexual risk behaviors. We are evaluating the effectiveness of the program primarily with confidential surveys of the participants before and after the program.

DETAILED DESCRIPTION:
Many adolescents in the U.S., even very young adolescents, are engaging in sexual risk behaviors that put them at risk for sexually transmitted diseases (STDs) and unintended pregnancy. Studies show that parents can play a significant role in promoting healthy sexual development and risk reduction among adolescents. Parenting approaches such as engaging in open and responsive communication, providing appropriate levels of supervision, and keeping involved in children's lives are associated with better adolescent outcomes. However, many parents are uncertain about how to talk with their adolescents about sex. Worksites provide an untapped but promising setting in which to reach parents to help them develop parenting and communication skills.

The UCLA/RAND Center for Adolescent Health Promotion has developed a worksite-based parenting program for parents of adolescents (grades 6-10) to improve parent-adolescent communication and reduce adolescent sexual risk behaviors. Specifically, the Center has developed Talking Parents, Healthy Teens for parents with adolescent children to teach communication skills as well as basic facts about sex and other important adolescent issues. The program aims to help parents understand adolescent development and the changes in adolescents' thoughts and feelings about sexual issues and other risk behaviors. It helps parents develop skills for discussing sensitive but important topics with their adolescents, and for teaching their adolescents decision-making and problem-solving skills. The program also emphasizes the importance of parents knowing what is going on in their adolescents' lives (often called parental monitoring). Although parents feel a need for help on such issues, they often tend to be too busy to attend ongoing programs. Therefore, we bring the program to them at their worksite. The program involves groups of about 12-15 parents who meet for an hour at lunch-time once a week for eight consecutive weeks. We serve a free lunch during the sessions.

We are evaluating the effectiveness of the Talking Parents, Healthy Teens program primarily with confidential surveys of the participants before and after the program. We also ask participants' adolescents (who are not in the parenting program) to fill out surveys as well. Among parents who initially express interest in the program, we randomize parents after they complete their baseline survey into an intervention group that takes the parenting program and a control group that does not. Both of these groups fill out confidential surveys over the course of several years. After the study has been conducted at a number of worksites, the research team will statistically compare survey answers for the two groups to see how well the program works. The results of the evaluation will be submitted for publication in academic journals.

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents in grades 6-10
* Parents must spend at least two days per week with their adolescents
* One parent per household/family

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1252 (Actual)
Dates: Start 2002-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Parent-child communication | 0, 3, 9, 15, 21, 27, 33, 39, & 45 months post-intervention

SECONDARY OUTCOMES:
Parenting behaviors | 0, 3, 9, 15, 21, 27, 33, 39, & 45 months post-intervention
Adolescent health behaviors | 0, 3, 9, 15, 21, 27, 33, 39, & 45 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Schuster, MD, PhD, Principal Investigator — RAND and UCLA
Locations (1):
- RAND, Santa Monica, California, United States

REFERENCES:
- [Background] Schuster MA, Eastman KL, Fielding JE, Rotheram-Borus MJ, Breslow L, Franzoi LL, Kanouse DE. Promoting adolescent health: worksite-based interventions with parents of adolescents. J Public Health Manag Pract. 2001 Mar;7(2):41-52. doi: 10.1097/00124784-200107020-00007. PMID 12174399
- [Background] Eastman KL, Corona R, Ryan GW, Warsofsky AL, Schuster MA. Worksite-based parenting programs to promote healthy adolescent sexual development: a qualitative study of feasibility and potential content. Perspect Sex Reprod Health. 2005 Jun;37(2):62-9. doi: 10.1363/psrh.37.062.05. PMID 15961359
- [Background] Eastman KL, Corona R, Schuster MA. Talking parents, healthy teens: a worksite-based program for parents to promote adolescent sexual health. Prev Chronic Dis. 2006 Oct;3(4):A126. Epub 2006 Sep 15. PMID 16978501
- [Result] Schuster MA, Corona R, Elliott MN, Kanouse DE, Eastman KL, Zhou AJ, Klein DJ. Evaluation of Talking Parents, Healthy Teens, a new worksite based parenting programme to promote parent-adolescent communication about sexual health: randomised controlled trial. BMJ. 2008 Jul 10;337:a308. doi: 10.1136/bmj.39609.657581.25. PMID 18617492